CLINICAL TRIAL: NCT03155282
Title: Diagnostic Accuracy of Spleen and Liver Stiffness Measurement by EUS-elastography, to Predict Portal Hypertension in Patients With Cirrhosis.
Brief Title: Utility of EUS-elastography to Predict Portal Hypertension
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: MAY 1-2017
Record Dates: First submitted 2017-05-13; First posted 2017-05-16 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhotic group: 30 patients with cirrhosis will be evaluated by EUS-E to measure liver and spleen stiffness. Different cirrhosis etiologies will be included like cirrhosis induces by alcohol, virus, autoimmune, nonalcoholic steatohepatitis (NASH), cryptogenic, primary sclerosing cholangitis and primary biliary cirrhosis. The cirrhotic status will be determinate by clinical, biochemical and/or imaging methods (abdominal ultrasound or CT scan).
  Interventions: Procedure: EUS-E to measure liver and spleen stiffness.
- Control group: 30 normal patients with no history of liver disease (negative hepatitis B virus and hepatitis C virus serology, insignificant alcohol intake, normal ultrasound and laboratory), in whom a EUS has to be performed to evaluate a esophageal or gastric subepithelial lesion, chronic pancreatitis, will be evaluated by EUS-E to measure liver and spleen stiffness.
  Interventions: Procedure: EUS-E to measure liver and spleen stiffness.

INTERVENTIONS:
Procedure: EUS-E to measure liver and spleen stiffness. — The EUS-E quantitative evaluation will be performed on the left hepatic lobe transgastrically. For the SR calculation, the area A will be manually selected including as much of hepatic tissue as possible and the area B will be selected on the red gastric mucosa. For the strain histogram measurement, the ROI selected will have a surface of 60 mm2. The same procedure will be repeated 10 times at different points on the left hepatic lobe and finally the mean SR and SH values will be calculated. The same sequence will be repeated to measure the spleen stiffness. Finally the azygos vein (AV) will be evaluated using EUS Doppler. The mean velocity and the AV diameter will be measure and the AV blood flow volume index (BFVI) will be calculated.

SUMMARY:
Patients with cirrhosis have structural and functional alterations of the liver. The progressive deposition of hepatic fibrosis is related to the subsequent development of portal hypertension (PH), and PH is associated with mayor complications including ascites, hepatic encephalopathy and development of gastroesophageal varices with a high risk of bleeding. Variceal bleeding is a medical emergency associated with a 6-week mortality rate of approximately 10-20%. Liver biopsy is the gold standard for the assessment of hepatic fibrosis, whereas the measurement of hepatic vein pressure gradient (HVPG) is the standard to evaluate PH and upper endoscopy (UE) is the method of choice to detect the presence and grade of gastroesophageal varices. The last two also estimates the risk of variceal bleeding. Unfortunately, clinical investigation of PH implies HVPG measurement or endoscopy for esophageal varices (EV) screening and grading. The first one is an invasive technique, mainly restricted to tertiary centers, that requires personal training, increased health care costs and patient discomfort. The UE, even though has demonstrated utility to predict HVPG (HVPG value ≥ 10 mmHg predicts the presence of EV and a value ≥ 12 mmHg is predictive for variceal bleeding), has been criticized of being subjective. Because of this, alternative test including elastographic techniques, have been develop to assess the severity of PH, the presence of EVs and the risk of variceal bleeding. Elastography is a technique used to measure tissue elasticity and stiffness in real time, by the application of slight compression using a transducer to the targeted tissue. The principle is that tissue compression produces deformation (strain) and that the strain is smaller in harder tissue as compared to softer tissue. Consequently, by measuring the tissue strain induced by compression, it is possible to estimate the tissue hardness. Fibroscan® (FS) (Echosens, París, Francia) uses the principle of one-dimension transient elastography (TE) for the assessment of tissue stiffness. It was used initially for liver stiffness measurement (LSM) and proved to be reliable for the diagnosis of liver cirrhosis and avoid liver biopsy in 90% of cases. Also LSM by TE accurately correlates with the severity of PH and the presence of esophageal varices.

DETAILED DESCRIPTION:
More recently, the use of Fibroscan for the spleen stiffness measurement (SSM) has become particularly attractive to assess. Previous studies have demonstrated that liver cirrhosis and PH generates some modifications in the spleen such as an increment in size, splenic blood flow, tissue hyperplasia, and fibrosis that determine an increase in the spleen's density and tissue stiffness that may be quantified by elastography. The SSM was found to be a valuable tool for assessing the degree of PH, the presence and severity of EVs and the risk of variceal bleeding among patients with cirrhosis. Moreover, spleen stiffness as compared with liver stiffness better represents the dynamic changes occurring in the advanced stages of cirrhosis and shows higher diagnostic performance in detecting esophageal varices.

Elastography can also be applied by endoscopic ultrasound (EUS-E). The EUS elastography allowed qualitative and quantitative evaluation. Qualitative elastography evaluates tissue elasticity by measuring the degree of deformation using a scale in the B-mode image of 1 to 255. This scale is represented by a color map (red- green-blue), wherein hard tissue is shown in dark blue, tissue with intermediate hardness in green, medium soft tissue in yellow, and soft tissue in red. There are two options for quantitative elastography and both are based on the qualitative EUS elastography data, the hue histogram and strain ratio. The hue histogram represents the overall elasticity within a manually selected area witch is the region of interest (ROI). The global hardness is being represent by a hue scale from 0 to 250, where 0 represents the hardest and 255 is the softest. The strain ratio (SR) analyzes the elastographic picture of the target lesion in relation to the surrounding tissues. Two different areas (A and B) are selected. Area A includes as much of the target lesion as possible without including the surrounding tissues. Area B is selected within a soft (red) reference area outside the target lesion, preferably the gut wall. The strain ratio is calculated as the quotient of B/A.

EUS is also a technique that has proved to be useful to evaluate cirrhotic patients in many aspects. It allows visualization of a greater part of the portal and portosystemic collateral circulation. It can be used to detect esophageal and gastric varices witch correlate with the presence and severity of liver disease and portal hypertension. It can be use to measure varices size. Large varices (≥ 5 mm) may be risk factors for variceal hemorrhage. It can visualize paramural collaterals and large vessels such as splenic, portal and azygos veins. Previous studies have found a significant increase in azygos vein diameter and blood-flow velocity in patients with varices when compared with control subjects. The evaluation of the azygos vein using EUS can ad useful information about the porto-systemic collateral circulation and could help to determine the treatment efficacy. It has been found a decrease in the azygos vein flow following terlipressin and somatostatin administration, band ligation or sclerotherapy in patients with portal hypertension. EUS can predict variceal recurrence after endoscopic therapy. Finally, cirrhosis causes dilation thoracic duct and thickening of gastric mucosa and submucosa that can be determinate by EUS.

MATERIAL AND METHODS

Study design: This is a prospective, observational, non-randomized and simple blind study, performed in a Tertiary Academic Center.

Setting: Ecuadorian Institute of Digestive Disease (IECED), Omni Hospital Academic Tertiary Center. Patients will be recruited from the gastroenterology unit (IECED), from January 2017 to June 2017. The study protocol and consent form has been approved by the Institutional Review Board and will be conducted according to the declaration of Helsinki. Written informed consent will be obtained from all participants.

Portal Hypertension determination: The HVPG will be determinate indirectly by upper endoscopy and clinical examination. A HVPG ≥ 10 mm Hg defines a clinically significant PH (CSPH) and will be determinate by the presence of EV on UE. On the other hand, a HVPG ≥ 12 mm Hg indicates a severe PH and will be determinate by the presence variceal bleeding on UE or ascites and hepatic encephalopathy.

The EUS procedure: The procedure will be performed under general anesthesia, with tracheal intubation, with the patient in supine position and in an endoscopy suite. All patients will be initially evaluated by upper endoscopy using a standard gastroscopy in order to avoid any contraindication and for gastro and esophageal varices assessment. Esophageal varices will be graded according to the Baveno VI consensus conference as follows: grade I, varices flattened by insufflation; grade II, varices non-confluent and protruding in the lumen despite insufflation; grade III, confluent varices not flattened by insufflation. Presence of red signs, fibrin plugs on the varices, and blood in the upper gastrointestinal tract will be also recorded. Gastric varices will be classified according to the classification of Sarin and Kumar. The EUS exam will be performed using a 3.8 mm working channel linear-array echoendoscopes (EG 3870UTK; Pentax, Hamburg, Germany), attached to an US console (Avius Hitachi, Tokyo, Japan). Two endoscopists (C.R.M, M.V) with experience in EUS-elastography will perform the procedures. The exam will start by evaluating the left hepatic lobe (the closer hepatic segment to the transducer) transgastrically using the conventional B-mode. Then the elastography software will be activated and the elastographic and B-mode images will be displayed simultaneously side by side, performing a real time qualitative evaluation of the hepatic tissue elasticity. The free movement of the endoscope tip, as well as sporadic motion of the tissues induced by respiratory or heart movements, determines lateral slippage of the target tissue. In order to avoid that, once the scope is located it will be fixed using the brakes. Images obtained with the application of strong pressure lead to wrong measures, so light pressure will be applied. The measurement will be considered adequate when the gastric mucosa is shown red. Once the transducer is correctly located the quantitative evaluation will be performed. For the SR calculation, the area A will be manually selected including as much of hepatic tissue as possible and the area B will be selected on the red gastric mucosa. For the strain histogram measurement, the ROI selected will have a surface of 60 mm2. Both values will be photographically recorded. The same procedure will be repeated 10 times at different points on the left hepatic lobe and finally the mean SR and SH values will be calculated. The procedure will continue by measuring the spleen stiffness. The transducer will be placed as close as possible to the spleen. Patients in whom the distance between the transducer and the spleen is more than 1.5 cm will be excluded from the analysis, but included in the intention to treat. The elastography software will be activated and the previously described sequence will be repeated. Ten measurements will be performed and the mean SR and SH values will be calculated. Finally the azygos vein (AV) will be scanned in all patients and evaluated using EUS Doppler. It will be scanned at a distance of 20-30 cm from the incisors with the EUS probe placed opposite to the posterior wall of the esophagus and to the right of the vertebral column. After the AV is found it will be followed until its arch. Measurements of the AV will be performed at a point just caudal to its arch, which drains into the superior vena cava. The angle of insonation will be less than 60º. The mean velocity (V mean cm/s) and the AV diameter (D) will be measure and the AV blood flow volume index (BFVI) will be calculated [BFVI (cm3 /s) = Vmean (cm/s) X D2 (cm2)]. The BFVI has been used before and it has been found to correlate with the blood-flow volume.

The Fibroscan procedure: In all patients, the liver stiffness measurements (LSM) will be assesses by transient elastography (TE) using the FibroScan® (FS) (Echosens, Paris, France). Spleen stiffness (SSM) measurement requires special software not approved by the National Administration of Food, Drugs and Technology. For the LSM, a previously described technique will be used. The patients will be in the supine position with arms in maximal abduction. The TE probe will be applied on the right lobe of the liver, via the intercostal spaces, in the right axillary midline and perpendicular to the plane of the skin. The results will be expressed in kilopascals (kPa). At least 10 LSM values will be carried out on each patient. The FS screen will show 3 parameters that have to be taken into account: the success rate calculated as the number of valid measurements divided by the number of total measurements, the median value calculated as average value of the 10 successful measurements and the interquartile range (IQR) calculated as the deviation of the total of valid measurements with respect to the median value. According to the manufacturer's recommendations and previous evidence, an interquartile range (IQR) ≥ 30% of the median value and success rate ≤ 60% will be considered incorrect and these patients will be excluded from the analysis but included in the intention to treat. LSM will be performed by two operators (H.P.L, J.O.A.), with more than 200 procedures performed each, blindly to the EUS-E results.

Statistical analysis: Baseline characteristics as age, gender will be compared between case and control group. Categorical variables will be assessed using Chi-square o Fisher Test and continuing variables with Student's t-test or Mann-Whitney Test. The relationships between the parameters will be characterized using the Spearman correlation coefficients and Pearson's correlation coefficient. The liver and spleen stiffness elastographic data will be expressed in kPa. All continuous variables will be expressed in mean ± standard deviation or median (range) as appropriate. The diagnostic performance of LSM and SSM by EUS elastography will be assessed using sensitivity (Se), specificity (Sp), positive predictive value (PPV), negative predictive value (NPV), accuracy, likelihood ratio (LR), Odds ratios (OR) with a 95% confidence intervals (CI) and receiver-operating characteristic (ROC) curves. Sensitivity analyses of patients under NSBB treatment prior elastography examination will be perform separately. Values of P < 0.05 will be considered significant. All the statistical analysis will be performed using SPSS software suite v.22. (Chicago, IL, USA).

Limitations: Since the examiner will have to choose the best EUS-E images from a dynamic sequence, a high examiner bias could be certainly favored. Selection of the ROI will be manually. In case of SH measure, the ROI will have in every case a 60 surface, but for SR measurement of the area A will have to include as tissue as possible with the possibility of differences between measurements. There are factors that have been described, especially with the use of the strain ratio that may influence the results of the elastography calculations. Examples are the presence of fluid (ascites, cysts, vessels) between the transducer and the ROI, the degree of compression by the transducer, the ROI diameter, the distance with the transducer, respiratory and cardiac movements, and the operator's experience. An attempt to reduce this factors will be apply, however they may not be completely eliminated in all the cases. The presence of ascites represents a more advanced stage of liver cirrhosis and a high risk of EV. However, the ascites limits the stiffness measurement by elastography and is considered and exclusion criteria. Therefore, most of the patients will be classified as Child-Pugh score A.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 - 80 years old.
* Who agree to participate in the study.
* Compensated liver cirrhotic patients (alcohol, virus, autoimmune, NASH, primary sclerosing cholangitis and primary biliary cirrhosis).

Exclusion Criteria:

* Moderate or severe perihepatic or perisplenic ascites. The presence of ascites limits the stiffness measurement.
* Acute and acute on chronic hepatitis. It aims to decrease the influence of inflammation in the elastography evaluation.
* Multiple focal liver lesions.
* Cholestatic liver disease and biliary obstruction.
* Failure to carry out liver TE by Fibroscan. Patients with an interquartile range (IQR) >30% of the median value and a success rate <60% will be excluded from the analysis but included in the intention to treat.
* Portal vein thrombosis.
* Esophageal, gastric, liver, spleen or pancreatic tumors that may impede to perform a correct EUS-E
* Cirrhotic patients with a recent episode of gastrointestinal bleeding or infection that may affect the hemodynamic flow.
* Splenectomy or history of partial splenic embolization.
* Pregnancy.
* Patient' s refusal to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with compensated liver cirrhosis will be recruit (cirrhosis induces by alcohol, virus, autoimmune, nonalcoholic steatohepatitis (NASH), cryptogenic, primary sclerosing cholangitis and primary biliary cirrhosis). Patients under β-blocker (BB) therapy will be evaluated independently. This medication acts by lowering portal pressure. Therefore, an effect on spleen stiffness cannot be ruled out. The control group will include normal patients with no history of liver disease, in whom a EUS has to be performed to evaluate a esophageal or gastric subepithelial lesion, chronic pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-10-29 (Actual)

PRIMARY OUTCOMES:
evaluate the accuracy of LSM and SSM by EUS-elastography (EUS-E) to assess PH in patients with liver cirrhosis and determinate if EUS-E can be used as a surrogate marker for PH. It also aims to find the optimal liver and spleen EUS-E values in predicting | 4 month
  The diagnostic performance of LSM and SSM by EUS elastography will be assessed using sensitivity (Se), specificity (Sp), positive predictive value (PPV), negative predictive value (NPV), accuracy, likelihood ratio (LR), Odds ratios (OR) with a 95% confidence intervals (CI) and receiver-operating characteristic (ROC) curves.

SECONDARY OUTCOMES:
correlation between LSM, using transient elastography (Fibroscan) and EUS-E. | 4 month
  Elastography values measured by EUS and Fibroscan will be correlated.
correlation between LSM and SSM by EUS-E and hemodynamic changes in the porto-systemic collateral circulation measure by an increase in azygos vein diameter and blood-flow velocity. | 4 month
  the azygos vein (AV) will be evaluated using EUS Doppler. The mean velocity (Vmean cm/s) and the AV diameter (D) will be measure and the AV blood flow volume index (BFVI) will be calculated [BFVI (cm3 /s) = Vmean (cm/s) X D2 (cm2)]. Finally BFVI will be correlated with LSM and SSM by EUS-E

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Madranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ophir J, Cespedes EI, Garra BS, et al. Elastography: ultrasound imaging of tissue strain and elastic modulus in vivo. Eur J Ultrasound 1996; 3:49-70.
- [Background] Bolognesi M, Boscato N. Spleen and liver cirrhosis: relationship between spleen enlargement and portal hypertension in patients with liver cirrhosis. In: Chen TM, ed. New Developments in Liver Cirrhosis Research. Hauppauge, NY: Nova Science Publishers, 2006; 49-67.
- [Background] Lucidarme D, Foucher J, Le Bail B, Costera L, Villars S, Forzy G, et al. The ratio interquartile range/median value of liver stiffness measurement is a key factor of accuracy of transient elastography (Fibroscans) for the diagnosis of liver fibrosis. Hepatology. 2007; 46: 318
- [Background] Robles-Medranda C. Gastroint Endosc. 2015; 79 (5): AB440
- [Result] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] Ripoll C, Groszmann R, Garcia-Tsao G, Grace N, Burroughs A, Planas R, Escorsell A, Garcia-Pagan JC, Makuch R, Patch D, Matloff DS, Bosch J; Portal Hypertension Collaborative Group. Hepatic venous pressure gradient predicts clinical decompensation in patients with compensated cirrhosis. Gastroenterology. 2007 Aug;133(2):481-8. doi: 10.1053/j.gastro.2007.05.024. Epub 2007 May 21. PMID 17681169
- [Result] Garcia-Tsao G, Bosch J. Management of varices and variceal hemorrhage in cirrhosis. N Engl J Med. 2010 Mar 4;362(9):823-32. doi: 10.1056/NEJMra0901512. No abstract available. PMID 20200386
- [Result] Bosch J, Garcia-Pagan JC, Berzigotti A, Abraldes JG. Measurement of portal pressure and its role in the management of chronic liver disease. Semin Liver Dis. 2006 Nov;26(4):348-62. doi: 10.1055/s-2006-951603. PMID 17051449
- [Result] Gao L, Parker KJ, Lerner RM, Levinson SF. Imaging of the elastic properties of tissue--a review. Ultrasound Med Biol. 1996;22(8):959-77. doi: 10.1016/s0301-5629(96)00120-2. PMID 9004420
- [Result] Castera L, Le Bail B, Roudot-Thoraval F, Bernard PH, Foucher J, Merrouche W, Couzigou P, de Ledinghen V. Early detection in routine clinical practice of cirrhosis and oesophageal varices in chronic hepatitis C: comparison of transient elastography (FibroScan) with standard laboratory tests and non-invasive scores. J Hepatol. 2009 Jan;50(1):59-68. doi: 10.1016/j.jhep.2008.08.018. Epub 2008 Oct 26. PMID 19013661
- [Result] Kazemi F, Kettaneh A, N'kontchou G, Pinto E, Ganne-Carrie N, Trinchet JC, Beaugrand M. Liver stiffness measurement selects patients with cirrhosis at risk of bearing large oesophageal varices. J Hepatol. 2006 Aug;45(2):230-5. doi: 10.1016/j.jhep.2006.04.006. Epub 2006 May 16. PMID 16797100
- [Result] Bureau C, Metivier S, Peron JM, Selves J, Robic MA, Gourraud PA, Rouquet O, Dupuis E, Alric L, Vinel JP. Transient elastography accurately predicts presence of significant portal hypertension in patients with chronic liver disease. Aliment Pharmacol Ther. 2008 Jun;27(12):1261-8. doi: 10.1111/j.1365-2036.2008.03701.x. Epub 2008 Apr 4. PMID 18397389
- [Result] Lemoine M, Katsahian S, Ziol M, Nahon P, Ganne-Carrie N, Kazemi F, Grando-Lemaire V, Trinchet JC, Beaugrand M. Liver stiffness measurement as a predictive tool of clinically significant portal hypertension in patients with compensated hepatitis C virus or alcohol-related cirrhosis. Aliment Pharmacol Ther. 2008 Nov 1;28(9):1102-10. doi: 10.1111/j.1365-2036.2008.03825.x. PMID 18691352
- [Result] Bolognesi M, Merkel C, Sacerdoti D, Nava V, Gatta A. Role of spleen enlargement in cirrhosis with portal hypertension. Dig Liver Dis. 2002 Feb;34(2):144-50. doi: 10.1016/s1590-8658(02)80246-8. PMID 11926560
- [Result] Kuddus RH, Nalesnik MA, Subbotin VM, Rao AS, Gandhi CR. Enhanced synthesis and reduced metabolism of endothelin-1 (ET-1) by hepatocytes--an important mechanism of increased endogenous levels of ET-1 in liver cirrhosis. J Hepatol. 2000 Nov;33(5):725-32. doi: 10.1016/s0168-8278(00)80302-5. PMID 11097479
- [Result] Colecchia A, Montrone L, Scaioli E, Bacchi-Reggiani ML, Colli A, Casazza G, Schiumerini R, Turco L, Di Biase AR, Mazzella G, Marzi L, Arena U, Pinzani M, Festi D. Measurement of spleen stiffness to evaluate portal hypertension and the presence of esophageal varices in patients with HCV-related cirrhosis. Gastroenterology. 2012 Sep;143(3):646-654. doi: 10.1053/j.gastro.2012.05.035. Epub 2012 May 27. PMID 22643348
- [Result] Calvaruso V, Bronte F, Conte E, Simone F, Craxi A, Di Marco V. Modified spleen stiffness measurement by transient elastography is associated with presence of large oesophageal varices in patients with compensated hepatitis C virus cirrhosis. J Viral Hepat. 2013 Dec;20(12):867-74. doi: 10.1111/jvh.12114. Epub 2013 Aug 12. PMID 24304456
- [Result] Colecchia A, Colli A, Casazza G, Mandolesi D, Schiumerini R, Reggiani LB, Marasco G, Taddia M, Lisotti A, Mazzella G, Di Biase AR, Golfieri R, Pinzani M, Festi D. Spleen stiffness measurement can predict clinical complications in compensated HCV-related cirrhosis: a prospective study. J Hepatol. 2014 Jun;60(6):1158-64. doi: 10.1016/j.jhep.2014.02.024. Epub 2014 Mar 6. PMID 24607624
- [Result] Stefanescu H, Grigorescu M, Lupsor M, Procopet B, Maniu A, Badea R. Spleen stiffness measurement using Fibroscan for the noninvasive assessment of esophageal varices in liver cirrhosis patients. J Gastroenterol Hepatol. 2011 Jan;26(1):164-70. doi: 10.1111/j.1440-1746.2010.06325.x. PMID 21175810
- [Result] Kim HY, Jin EH, Kim W, Lee JY, Woo H, Oh S, Seo JY, Oh HS, Chung KH, Jung YJ, Kim D, Kim BG, Lee KL. The Role of Spleen Stiffness in Determining the Severity and Bleeding Risk of Esophageal Varices in Cirrhotic Patients. Medicine (Baltimore). 2015 Jun;94(24):e1031. doi: 10.1097/MD.0000000000001031. PMID 26091449
- [Result] Giunta M, Conte D, Fraquelli M. Role of spleen elastography in patients with chronic liver diseases. World J Gastroenterol. 2016 Sep 21;22(35):7857-67. doi: 10.3748/wjg.v22.i35.7857. PMID 27672283
- [Result] Iglesias-Garcia J, Lindkvist B, Larino-Noia J, Dominguez-Munoz JE. Endoscopic ultrasound elastography. Endosc Ultrasound. 2012 Apr;1(1):8-16. doi: 10.7178/eus.01.003. PMID 24949330
- [Result] Faigel DO, Rosen HR, Sasaki A, Flora K, Benner K. EUS in cirrhotic patients with and without prior variceal hemorrhage in comparison with noncirrhotic control subjects. Gastrointest Endosc. 2000 Oct;52(4):455-62. doi: 10.1067/mge.2000.107297. PMID 11023560
- [Result] Salama ZA, Kassem AM, Giovannini M, Hunter MS. Endoscopic ultrasonographic study of the azygos vein in patients with varices. Endoscopy. 1997 Oct;29(8):748-50. doi: 10.1055/s-2007-1004301. PMID 9427495
- [Result] Caletti G, Brocchi E, Baraldini M, Ferrari A, Gibilaro M, Barbara L. Assessment of portal hypertension by endoscopic ultrasonography. Gastrointest Endosc. 1990 Mar-Apr;36(2 Suppl):S21-7. doi: 10.1016/s0016-5107(90)71011-5. PMID 2184082
- [Result] Kassem AM, Salama ZA, Zakaria MS, Hassaballah M, Hunter MS. Endoscopic ultrasonographic study of the azygos vein before and after endoscopic obliteration of esophagogastric varices by injection sclerotherapy. Endoscopy. 2000 Aug;32(8):630-4. doi: 10.1055/s-2000-9018. PMID 10935792
- [Result] Lee YT, Sung JJ, Yung MY, Yu AL, Chung SC. Use of color Doppler EUS in assessing azygos blood flow for patients with portal hypertension. Gastrointest Endosc. 1999 Jul;50(1):47-52. doi: 10.1016/s0016-5107(99)70343-3. PMID 10385721
- [Result] Yokoyama M, Shijo H, Ota K, Kubara K, Kokawa H, Kim T, Akiyoshi N, Okumura M, Inoue K. Systemic hemodynamics and serum nitrate levels in patients undergoing endoscopic variceal ligation. Hepatology. 1996 Jul;24(1):47-52. doi: 10.1053/jhep.1996.v24.pm0008707281.
- [Result] Sugano S, Yamamoto K, Takamura N, Momiyama K, Watanabe M, Ishii K. Azygos venous blood flow while fasting, postprandially, and after endoscopic variceal ligation, measured by magnetic resonance imaging. J Gastroenterol. 1999 Jun;34(3):310-4. doi: 10.1007/s005350050266. PMID 10433004
- [Result] Yokoyama M, Shijo H, Ota K, Kubara K, Kokawa H, Kim T, Akiyoshi N, Tokumitsu H, Okumura M. Effects of endoscopic variceal sclerotherapy on azygos vein blood flow and systemic haemodynamics. J Gastroenterol Hepatol. 1996 Aug;11(8):780-5. doi: 10.1111/j.1440-1746.1996.tb00332.x. PMID 8872779
- [Result] Hammoud GM, Ibdah JA. Utility of endoscopic ultrasound in patients with portal hypertension. World J Gastroenterol. 2014 Oct 21;20(39):14230-6. doi: 10.3748/wjg.v20.i39.14230. PMID 25339809
- [Result] Castera L, Pinzani M, Bosch J. Non invasive evaluation of portal hypertension using transient elastography. J Hepatol. 2012 Mar;56(3):696-703. doi: 10.1016/j.jhep.2011.07.005. Epub 2011 Jul 20. PMID 21767510
- [Result] Sarin SK, Kumar A. Gastric varices: profile, classification, and management. Am J Gastroenterol. 1989 Oct;84(10):1244-9. PMID 2679046
- [Result] Frey H. [Realtime elastography. A new ultrasound procedure for the reconstruction of tissue elasticity]. Radiologe. 2003 Oct;43(10):850-5. doi: 10.1007/s00117-003-0943-2. German. PMID 14605701
- [Result] Giovannini M, Hookey LC, Bories E, Pesenti C, Monges G, Delpero JR. Endoscopic ultrasound elastography: the first step towards virtual biopsy? Preliminary results in 49 patients. Endoscopy. 2006 Apr;38(4):344-8. doi: 10.1055/s-2006-925158. PMID 16680632
- [Result] Ziol M, Handra-Luca A, Kettaneh A, Christidis C, Mal F, Kazemi F, de Ledinghen V, Marcellin P, Dhumeaux D, Trinchet JC, Beaugrand M. Noninvasive assessment of liver fibrosis by measurement of stiffness in patients with chronic hepatitis C. Hepatology. 2005 Jan;41(1):48-54. doi: 10.1002/hep.20506. PMID 15690481
- [Result] Castera L, Forns X, Alberti A. Non-invasive evaluation of liver fibrosis using transient elastography. J Hepatol. 2008 May;48(5):835-47. doi: 10.1016/j.jhep.2008.02.008. Epub 2008 Feb 26. PMID 18334275
- [Result] Kettaneh A, Marcellin P, Douvin C, Poupon R, Ziol M, Beaugrand M, de Ledinghen V. Features associated with success rate and performance of FibroScan measurements for the diagnosis of cirrhosis in HCV patients: a prospective study of 935 patients. J Hepatol. 2007 Apr;46(4):628-34. doi: 10.1016/j.jhep.2006.11.010. Epub 2006 Dec 12. PMID 17258346
- [Result] Boursier J, Zarski JP, de Ledinghen V, Rousselet MC, Sturm N, Lebail B, Fouchard-Hubert I, Gallois Y, Oberti F, Bertrais S, Cales P; Multicentric Group from ANRS/HC/EP23 FIBROSTAR Studies. Determination of reliability criteria for liver stiffness evaluation by transient elastography. Hepatology. 2013 Mar;57(3):1182-91. doi: 10.1002/hep.25993. Epub 2013 Feb 4. PMID 22899556
- [Result] Sandrin L, Fourquet B, Hasquenoph JM, Yon S, Fournier C, Mal F, Christidis C, Ziol M, Poulet B, Kazemi F, Beaugrand M, Palau R. Transient elastography: a new noninvasive method for assessment of hepatic fibrosis. Ultrasound Med Biol. 2003 Dec;29(12):1705-13. doi: 10.1016/j.ultrasmedbio.2003.07.001. PMID 14698338
- [Result] Dawwas MF, Taha H, Leeds JS, Nayar MK, Oppong KW. Diagnostic accuracy of quantitative EUS elastography for discriminating malignant from benign solid pancreatic masses: a prospective, single-center study. Gastrointest Endosc. 2012 Nov;76(5):953-61. doi: 10.1016/j.gie.2012.05.034. Epub 2012 Jul 31. PMID 22854060
- [Derived] Termite F, Borrelli de Andreis F, Liguori A, Gasbarrini A, Attili F, Spada C, Miele L. The Role of Endoscopic Ultrasound in Assessing Portal Hypertension: A State-of-the-Art Literature Review and Evolving Perspectives. Liver Int. 2025 Apr;45(4):e16176. doi: 10.1111/liv.16176. Epub 2024 Nov 27. PMID 39601324